CLINICAL TRIAL: NCT00112359
Title: A Phase 3, Double-Blind, Multicenter, Multinational, Randomized, Placebo-Controlled Trial Evaluating Aztreonam Lysinate for Inhalation in Cystic Fibrosis Patients With Pulmonary Pseudomonas Aeruginosa (AIR-CF1)
Brief Title: International Safety and Efficacy Study of Aztreonam for Inhalation Solution (AZLI) in Cystic Fibrosis Patients With P. Aeruginosa
Acronym: AIR-CF1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Mark Bresnik, MD, Director, Clinical Research, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-AI-007
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa; Pulmonary Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo three times a day (TID) (Placebo Comparator)
  Interventions: Drug: Placebo three times a day (TID)
- AZLI 75 mg three times a day (TID) (Experimental)
  Interventions: Drug: AZLI 75 mg three times a day (TID)

INTERVENTIONS:
Drug: AZLI 75 mg three times a day (TID)
  Arms: AZLI 75 mg three times a day (TID)
Drug: Placebo three times a day (TID)
  Arms: Placebo three times a day (TID)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of a 28-day course of aztreonam for inhalation solution (AZLI) in patients with cystic fibrosis (CF) and lung infection due to Pseudomonas aeruginosa (PA).

DETAILED DESCRIPTION:
CF patients often have lung infections that occur repeatedly or worsen over time. The lung infections are often caused by a bacteria called Pseudomonas aeruginosa (PA). Treatment with antibiotics can stop or slow down the growth of the bacteria. The antibiotics may be given by mouth, intravenously (IV), or by inhalation as a mist. The purpose of this study was to evaluate the safety and efficacy of AZLI, an investigational formulation of the antibiotic aztreonam and administered TID using the PARI eFlow® electronic nebulizer, in CF patients with PA.

In this study, participant eligibility was assessed at a screening visit 7 to 14 days prior to the baseline visit (Day 0). Those participants who continued to meet eligibility criteria at Day 0 were randomized and began a 28-day course of blinded study treatment (AZLI TID or placebo TID). Participants returned for clinic visits at Day 14, an end of treatment visit at Day 28, and a follow-up visit 14 days after the last dose of study drug (Day 42).

ELIGIBILITY:
Inclusion Criteria:

* Documentation of CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

  * Sweat chloride greater than or equal to 60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT);
  * Two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene; or
  * Abnormal nasal potential difference.
* PA present in expectorated sputum or throat swab culture at Screening.
* FEV1 between (and including) 25% and 75% predicted at Screening.
* Negative pregnancy test at Screening.
* Ability to perform reproducible pulmonary function tests.
* Arterial oxygen saturation (SaO2) greater than or equal to 90% on room air at Screening.
* Ability to provide written informed consent.

Exclusion Criteria:

* Administration of antipseudomonal antibiotics by inhalation, IV, or oral routes (including azithromycin) within 14 days of Screening.
* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone/day or 20 mg prednisone every other day.
* History of sputum or throat swab culture yielding Burkholderia cepacia in the previous 2 years.
* History of daily continuous oxygen supplementation or requirement for more than 2 liters/minute at night.
* Administration of any investigational drug or use of any investigational device within 28 days of Screening and within 6 half-lives of the investigational drug (whichever was longer).
* Known local or systemic hypersensitivity to monobactam antibiotics.
* Inability to tolerate short-acting bronchodilator use at least three times daily.
* Changes in protocol-permitted antimicrobial, bronchodilator, anti-inflammatory, or corticosteroid medications within 7 days prior to Screening or between Screening and the next visit.
* Changes in physiotherapy technique or schedule within 7 days prior to Screening or between Screening and the next visit.
* History of lung transplantation.
* A chest x-ray indicating abnormal findings at Screening or within the previous 90 days.
* Abnormal renal or hepatic function at Screening.
* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would have interfered with participant treatment, assessment, or compliance with the protocol.
* Use of aerosolized hypertonic saline (except for sputum induction) during the 14 days preceding Visit 1.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, MD, Study Director — Corus Pharma, Inc.
Locations (53):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pediatric Breathing Disorders Clinic, Anchorage, Alaska
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital, Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Capital Allergy and Respiratory Disease Center, Sacramento, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Nemours Children's Clinic, Orlando, Orlando, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital / Northwestern University, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Via Christi - St. Francis Regional Medical Center, Wichita, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Central Maine Pulmonary Associates, Auburn, Maine
  - University of Michigan, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - Children's Lung Specialists, Las Vegas, Nevada
  - St. Barnabas Healthcare System, Livingston, New Jersey
  - Albany Medical College, Albany, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Pediatric Pulmonary Associates, South Carolina, Columbia, South Carolina
  - Baylor Martha Foster Lung Care Center, Dallas, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Naval Medical Center, Portsmouth, Virginia
  - Pediatric Pulmonary Center/Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (7):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (5):
  - Capital Health and the Governors of the University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Brian Lyttle Professional Corporation, London, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Auckland District Health Board, Auckland, New Zealand

REFERENCES:
- [Derived] Retsch-Bogart GZ, Quittner AL, Gibson RL, Oermann CM, McCoy KS, Montgomery AB, Cooper PJ. Efficacy and safety of inhaled aztreonam lysine for airway pseudomonas in cystic fibrosis. Chest. 2009 May;135(5):1223-1232. doi: 10.1378/chest.08-1421. PMID 19420195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 3, double-blind, multicenter, multinational, randomized, placebo-controlled trial evaluating AZLI in patients with CF and PA. Participants were enrolled at 53 sites total: 40 in United States, 5 in Canada, 7 in Australia, and 1 in New Zealand. Date of first enrollment was 10 Jun 2005, and date of last participant follow-up was 3 Apr 2007.
Pre-assignment Details: Planned study size was 140 participants to be randomized in a 1:1 ratio to AZLI or placebo TID, with 166 actually randomized (83 AZLI, 83 placebo). However, two participants did not receive a dose of drug, and one participant randomized to receive AZLI received placebo in error. Thus, 80 participants received AZLI and 84 received placebo.
Groups:
- Placebo TID: Placebo (5 mg/mL lactose when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.5, and osmolality 200 to 400 mOsmol/kg). Placebo was self-administered three times a day by inhalation using the investigational nebulizer.
- 75 mg AZLI TID: AZLI (75 mg/mL aztreonam lysine when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.0, and osmolality 300 to 550 mOsmol/kg). AZLI was self-administered by inhalation three times a day using the investigational nebulizer.
Period: Overall Study
Arm/Group | Placebo TID | 75 mg AZLI TID
Started | 84 | 80
Completed | 57 | 67
Not Completed | 27 | 13
Not completed — Unrelated adverse event | 16 | 8
Not completed — Trial drug intolerance (adverse event) | 2 | 0
Not completed — Related adverse event | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Personal/administrative | 1 | 1
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo TID | 75 mg AZLI TID | Total
Number analyzed (Participants) | 84 | 80 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 21 | 37
  Between 18 and 65 years | 66 | 59 | 125
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 31.7 (14.8) | 27.4 (12.8) | 29.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 71
  Male | 45 | 48 | 93
Region of Enrollment [Number; unit: participants]
  North America | 63 | 62 | 125
  Australia | 21 | 18 | 39
Disease severity based on forced expiratory volume in 1 second (FEV1) % predicted [Number; unit: participants] — FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height. This baseline measure indicates the number of subjects with FEV1 greater than 50% and less than or equal to 50% of the predicted value based on age, gender, and height at screening.
  participants
    Disease severity: FEV1 > 50% predicted | 54 | 50 | 104
    Disease severity: FEV1 <= 50% predicted | 30 | 30 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Change in CFQ-R RSS Score
Description: The CFQ-R was administered at baseline and every visit thereafter. The endpoint was change in respiratory symptoms from baseline, assessed with the CFQ-R RSS (range of scores: 0-100; higher scores indicate fewer symptoms).
Time Frame: Day 0 to Day 14
Population: ITT population: participants randomized to treatment who received at least part of 1 dose of study drug. Participants summarized by actual treatment received. Missing baseline data not imputed. Missing post-baseline data imputed using worst-case value for withdrawals due to AE or study drug intolerance. All other missing data: LOCF method used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 83 | 80
units on a scale | 0.976 (1.624) | 7.007 (1.647)
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in CFQ-R RSS score at Day 14; Test type: Superiority or Other; p = 0.0006, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included treatment, baseline CFQ-R RSS, and disease severity (FEV1 >50% or <=50% pred.). Treatment differences: AZLI-placebo; Mean Difference (Final Values) = 7.98, 95% CI 2-sided [3.50 to 12.47]

2. Secondary Outcome: Change in CFQ-R RSS Score
Description: as for outcome 1
Time Frame: Day 0 to Day 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 83 | 80
units on a scale | -5.711 (1.849) | 0.618 (1.875)
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in CFQ-R RSS score at Day 42; Test type: Superiority or Other; p = 0.0154, ANCOVA — No adjustments were made for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.33, 95% CI 2-sided [1.22 to 11.43]

3. Other Pre Specified Outcome: Number of Participants With Other Pathogens Present
Description: Sputum samples were collected at all visits for quantitative and qualitative culture for Staphylococcus aureus, Burkholderia cepacia, Stenotrophomonas maltophilia, Achromobacter xylosoxidans.
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). Participants were summarized by the actual treatment received. No imputation methods were used for the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 81 | 74
participants
  Staphylococcus aureus - Day 0 | 30 | 37
  Staphylococcus aureus - Day 28 | 31 | 35
  Burkholderia cepacia - Day 0 | 0 | 1
  Burkholderia cepacia - Day 28 | 0 | 0
  Stenotrophomonas maltophilia - Day 0 | 4 | 1
  Stenotrophomonas maltophilia - Day 28 | 2 | 2
  Achromobacter xylosoxidans - Day 0 | 5 | 1
  Achromobacter xylosoxidans - Day 28 | 7 | 1

4. Other Pre Specified Outcome: Minimum Inhibitory Concentration of Aztreonam Inhibiting 50% (MIC50) and 90% (MIC90) of All PA Isolates (μg/mL)
Description: PA isolates from sputum samples (collected at all visits) were assessed for their susceptibility to aztreonam.
  MIC50 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 50% of isolates from a particular organism).
  MIC90 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 90% of isolates from a particular organism).
  MIC50 and MIC90 values are single measurements for the entire population and not measured on a per-participant basis.
Time Frame: Day 0
Population: as for outcome 3
Measure: Number; unit: μg/mL
Units Other Than Participants: PA isolates
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 84 | 80
Number analyzed (PA isolates) | 140 | 128
μg/mL
  Day 0 MIC50 | 2 | 4
  Day 0 MIC90 | 64 | 128

5. Secondary Outcome: Percent Change in FEV1 (L)
Description: Spirometry was performed according to American Thoracic Society (ATS) guidelines at each visit. The percent change from baseline in forced expiratory volume (liters) in one second (FEV1) was determined at Day 28.
Time Frame: Day 0 to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change in FEV1 (L)
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 84 | 80
Percent change in FEV1 (L) | -2.408 (1.466) | 7.886 (1.481)
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in percent change in FEV1 at Day 28; Test type: Superiority or Other; p < 0.0001, ANCOVA — Analysis based on two-sided test with an 0.025 a priori threshold for statistical significance as part of the methods used to control the family-wise type 1 error; ANCOVA model included treatment, disease severity (FEV1 >50% or <=50% pred.), and Day 0 FEV1. Treatment differences: AZLI-placebo; Median Difference (Final Values) = 10.294, 95% CI 2-sided [6.288 to 14.299]

6. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa (PA) Log10 Colony Forming Units (CFU) Per Gram of Sputum
Description: Sputum samples were collected at all participant visits of the study for analysis of microbiology endpoints. Sputum samples were processed for qualitative and quantitative culture of PA (each morphotype). Due to the skewness of the distribution of CFU data, the data were transformed using the base 10 logarithm, in an attempt to normalize the data and allow for parametric tests, before calculating changes. To account for zero values, 1 was added to each CFU measurement before being transformed. Any CFU data values where PA was not isolated from a valid culture were set to zero.
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants randomized to treatment who received at least part of 1 dose of study drug). Participants were summarized by the actual treatment received. No imputation methods were used for the analysis.
Measure: Least Squares Mean (Standard Error); unit: Log10 PA CFUs/gram of sputum
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 61 | 53
Log10 PA CFUs/gram of sputum | 0.069 (0.231) | -1.384 (0.247)
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change in log10 PA CFUs in sputum at Day 28; Test type: Superiority or Other; p < 0.0001, ANCOVA — Analysis based on 2-sided test with an 0.025 a priori threshold for statistical significance as part of methods used to control family-wise type 1 error; ANCOVA model included terms for treatment and disease severity (FEV1 >50% or <=50% pred.). Treatment differences calculated as AZLI-placebo; Mean Difference (Final Values) = -1.453, 95% CI 2-sided [-2.115 to -0.791]

7. Secondary Outcome: Number of Participants Receiving Intravenous (IV) or Inhaled Antipseudomonal Antibiotics Other Than Trial Drug
Description: Use of IV and inhaled antipseudomonal antibiotics was compiled from data recorded on the Concomitant Medications eCRF.
Time Frame: Day 0 to Day 42
Population: Analysis based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). Participants were summarized by the actual treatment received.
Measure: Number; unit: participants
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 84 | 80
participants | 19 | 12
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in number of participants using additional (nonprotocol-specified) antipseudomonal antibiotics during study; Test type: Superiority or Other; p = 0.2364, Fisher Exact — [p-value comment as in outcome 6, analysis 1]; Comparison by treatment for proportion of subjects using additional (nonprotocol-specified) antipseudomonal antibiotics at least once during study

8. Primary Outcome: Change in CFQ-R Respiratory Symptoms Scale (RSS) Score
Description: The CFQ-R was administered at baseline and every visit thereafter. The endpoint was change in respiratory symptoms from baseline, assessed with the CFQ-R respiratory symptoms scale (RSS; range of scores: 0-100; higher scores indicate fewer symptoms).
Time Frame: Day 0 to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 83 | 80
units on a scale | -2.63 (1.95) | 7.08 (1.98)
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in CFQ-R RSS score at Day 28. A sample size of 70 participants per treatment group provided approximately 77% power to detect an 8-point difference in CFQ-R RSS score between treatment groups, assuming a standard deviation (SD) of 20 and a Type I error rate of 0.05; Test type: Superiority or Other; p = 0.0005, ANCOVA — Primary endpoint analysis based on 2-sided test with an 0.05 a priori threshold for statistical significance. A gate-keeping procedure to control family-wise Type 1 error was established a priori for primary and key secondary endpoints; ANCOVA model includes treatment, baseline CFQ-R RSS, and disease severity (FEV1 >50% or <=50% pred.). Treatment differences: AZLI-placebo; Mean Difference (Final Values) = 9.71, 95% CI 2-sided [4.31 to 15.11]

9. Secondary Outcome: Number of Participants Hospitalized at Least Once Between Day 0 and Day 42
Description: Details of all hospitalizations, including the dates of admission and discharge, were recorded on the SAE eCRF.
Time Frame: Day 0 to Day 42
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 84 | 80
participants | 12 | 4
Statistical Analysis 1: Comparison: Placebo TID vs 75 mg AZLI TID; Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in number of participants hospitalized at least once during the study; Test type: Superiority or Other; p = 0.0640, Fisher Exact — No adjustments were made for multiple comparisons; Comparison by treatment group for proportion of participants hospitalized at least once between Day 0 and Day 42 (or 14 days after last study dose)

10. Other Pre Specified Outcome: Minimum Inhibitory Concentration of Aztreonam Inhibiting 50% (MIC50) and 90% (MIC90) of All PA Isolates (μg/mL)
Description: as for outcome 4
Time Frame: Day 28
Population: as for outcome 3
Measure: Number; unit: μg/mL
Units Other Than Participants: PA isolates
Arm/Group | Placebo TID | 75 mg AZLI TID
Number analyzed (Participants) | 84 | 80
Number analyzed (PA isolates) | 116 | 102
μg/mL
  Day 28 MIC50 | 2 | 8
  Day 28 MIC90 | 64 | 128

ADVERSE EVENTS:
Time Frame: AEs that first occurred or worsened after the first dose of study drug through 30 days after the last dose are summarized.
Description: An AE was any physical or clinical worsening in symptoms or disease (including clinically significant change in lab values) experienced by participant at any time during the study, whether or not the event was considered related to study participation or study procedures.
  Participants were only counted once within an SOC and preferred term.
Arm/Group | Placebo TID | 75 mg AZLI TID
Serious Adverse Events (participants affected / at risk) | 12/84 | 5/80
Other Adverse Events (participants affected / at risk) | 67/84 | 63/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo TID (N=84) | 75 mg AZLI TID (N=80)
Asthenia (General disorders) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Intercostal retraction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Oxygen saturation decreased (Investigations) | 2 | 0
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pulmonary function test decreased (Investigations) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo TID (N=84) | 75 mg AZLI TID (N=80)
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 38
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Fatigue (General disorders) | 6 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Headache (Nervous system disorders) | 10 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 23 | 12
Pulmonary function test decreased (Investigations) | 5 | 3
Pyrexia (General disorders) | 6 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and investigator may publish or present the results of the trial generated there with prior written consent of Gilead; or 2 years after the trial has ended at all institutions. Proposed publications/target venue must go to Gilead 30 days (manuscripts) or 15 days (abstracts/presentations) prior. Any Gilead confidential information in the document(s) must be deleted, or if requested publication delayed for up to 45 days to permit Gilead to obtain intellectual property protection.